CLINICAL TRIAL: NCT04658771
Title: Pivotal / Phase II Clinical Trial of Magnetic Resonance-Guided Focused Ultrasound (MR-HIFU) Treatment of Painful Osteoid Osteoma in Children and Young Adults
Brief Title: MR-HIFU Treatment of Painful Osteoid Osteoma
Status: Active, not recruiting | Phase: Phase 2 | Type: Interventional
Sponsor: Children's National Research Institute (Other)
Responsible Party: Principal Investigator, Karun Sharma MD, Director of Interventional Radiology, Children's National Research Institute
Allocation: Not Applicable | Model: Single Group | Masking: None | Purpose: Treatment
Other Study IDs: HIFU OO Phase II
Record Dates: First submitted 2020-11-13; First posted 2020-12-08 (Actual); Last update posted 2025-07-11 (Actual); Status verified 2025-07

CONDITIONS: Osteoid Osteoma
MeSH Terms: conditions — Osteoma, Osteoid

STUDY DESIGN:
Oversight: Data Monitoring Committee: Yes | FDA-regulated Drug: No | FDA-regulated Device: Yes

ARMS (1):
- All patients (Experimental): Patients will undergo MR-HIFU ablation procedure of OO under general anesthesia. Patients will be monitored for disease status and adverse events for 12 months following procedure. Patients with incomplete or partial response at 28 days after MR-HIFU will be permitted a second MR-HIFU procedure.
  If there is still incomplete pain relief without medication use by 28 days following the second MR-HIFU treatment, patients will be offered standard of care treatment with RFA and followed for one year.
  Interventions: Device: MR-HIFU treatment

INTERVENTIONS:
Device: MR-HIFU treatment — MR-HIFU is an innovative technology that allows for non-invasive thermal ablation of tissues and tumors by integrating an external high intensity focused ultrasound (HIFU) transducer with a conventional MRI scanner.
  The focused ultrasound transducer is placed outside of the body and generates and focuses acoustic energy to heat tumors or other pre-defined focal regions of tissues inside the body. Because the acoustic energy is precisely focused over tiny areas of tissue, potential thermal injury to surrounding tissues is minimal. Cell death inside the selected treatment area occurs via coagulative necrosis while avoiding injury to intervening and adjacent tissues.

SUMMARY:
To determine treatment safety and efficacy of MR-HIFU ablation of painful Osteoid Osteoma (OO) in children and young adults.

DETAILED DESCRIPTION:
Osteoid Osteoma (OO) is a benign, but painful, bone tumor commonly occurring in children and young adults. Definitive treatment options are CT-guided radiofrequency ablation (RFA) and less commonly, open surgical resection. RFA is less invasive than surgery, but it still requires drilling from the skin through muscle and bone. It also exposes the patient and operator to ionizing radiation.

Magnetic Resonance guided High Intensity Focused Ultrasound (MR-HIFU) provides precise and controlled delivery of focused ultrasound energy inside a lesion using an external applicator, without any incisions or drilling. MR-HIFU has been successfully used to treat painful bone metastases in adult clinical trials. Several recent reports, including two publications from our group, show that MR-HIFU is a feasible and safe treatment for OO.

MR-HIFU ablation of OO may provide a better alternative to surgical resection or RFA as it is completely non-invasive and does not require ionizing radiation. These two qualities of MR-HIFU are especially beneficial in growing children and young adults. Furthermore, MR-HIFU OO ablation is quick, with expected total procedure time of less than two hours. Such short treatments offer additional safety benefits from reduced anesthesia / sedation requirement compared to surgery and RFA.

The investigator's group has performed the first pilot clinical trial in the U.S. to evaluate MR-HIFU treatment for painful osteoid osteoma (PI: K.V. Sharma, NCT02349971). This trial shows that MR-HIFU ablation is feasible, well tolerated, and can be safely performed in a pediatric cohort. Based on these results, the investigators propose a pivotal clinical trial designed to evaluate treatment efficacy as the next logical step required for clinical translation. The investigators hypothesize that noninvasive and radiation-free MR-HIFU ablation for osteoid osteoma will be a clinically effective treatment, with success rate comparable to that currently reported for RFA.

ELIGIBILITY:
Inclusion Criteria:

* Age ≤30 years.
* Diagnosis of OO: All patients diagnosed with painful OO based on characteristic clinical history of pain relieved with NSAID medications AND confirmatory imaging findings characteristic of OO on CT and/or MRI scans.
* Location of OO: eligible lesions must be located in a bone with acoustic accessibility and within the normal safety margins of MR-HIFU, as specified in the instructions for use.
* Prior therapy: Patients with prior unsuccessful treatments including CT-RFA and/or surgical resection are eligible for enrollment.
* Patients < 18 years old must be accompanied by a legal guardian at the time of recruitment.
* Laboratory:

  * Complete Blood Count (CBC) values within acceptable range for safe administration of anesthesia. Hemoglobin > 9 g/dL.
  * PT, PTT and INR < 1.5 x ULN (including patients on prophylactic anticoagulation)
  * Basic metabolic panel (BMP) and/or Complete metabolic panel (CMP) values within acceptable range for safe administration of anesthesia.
  * Adequate renal function: Age-adjusted normal serum creatinine (see table below) OR a creatinine clearance ≥60 mL/min/1.73 m2 for safe contrast administration
  * Adequate pulmonary function: Defined as no dyspnea at rest, and a pulse oximetry >94% on room air.

Exclusion Criteria:

* Diagnosis of bone lesion other than OO in the judgement of the Principal Investigator.
* Clinically significant unrelated systemic illness, such as serious infections, hepatic, renal or other organ dysfunction, which would compromise the patient's ability to tolerate the general anesthetic required for the procedure in the judgment of the Principal Investigator.
* Implant, prosthesis or scar tissue that would interfere with a safe completion of MR-HIFU. ablation in the judgement of the Principal Investigator.
* Treatment area nidus <1 cm from a major nerve, spinal canal, bladder, or bowel.
* Target <1 cm of growth plate (physis).
* Lesion in the skull.
* Lesion in the vertebral body.
* Inability to undergo MRI and/or contraindication for MRI.
* Inability to tolerate stationary position during MR-HIFU.
* Patients currently receiving any investigational agents.

Ages: 0 Years to 30 Years | Sex: All | Healthy Volunteers: No
Age Groups: Child, Adult
Enrollment: 30 (Estimated)
Dates: Start 2021-01-28 (Actual); Primary Completion 2024-06-11 (Actual); Study Completion 2025-12-30 (Estimated)

PRIMARY OUTCOMES:
Number of participants with treatment-related adverse events as assessed by the Common Terminology Criteria for Adverse Events (CTCAE) v.5 | 12 months
  CTCAE v.5 will be used
Pain relief as assessed by pain medication usage | 12 months
  The patient pain and medication diary will be used
Pain relief as assessed using the Visual Analog Scale (VAS) | 12 months
  The VAS is a continuous numerical pain scale ranging from 0 (no pain) to 10 (worst possible pain)
Pain relief as assessed by using the PROMIS Pain Interference short form | 12 months
  The PROMIS Pain Interference Short Form consists of 8 questions on pain. Each question will be rated from 0 (never), 1 (almost never), 2 (sometimes), 3 (often), and 4 (almost always)
Quality of life as assessed by using the Pediatric Quality of Life Inventory (PedsQL) v4.0 | 12 months
  The PedsQL is a 23-item, 4 scale, and 2 domain instrument measuring physical, social, emotional, and cognitive well-being. Each question will be rated from 0 (never) to 4 (almost always)
Quality of life as assessed by using the Symptom Distress Scale (SDS) | 12 months
  SDS is a 10-item Likert format instrument that measures symptom intensity and distress. Each question will be rated from 1 (no problems in the area) to 5 (worst problems in this area)

SECONDARY OUTCOMES:
Number of participants with change in nidus size (mm) as assessed via MRI | 12 months
  Number of participants with change in nidus size (mm) as assessed via MRI
Number of participants with change in nidus vascularity as assessed via MRI | 12 months
  Number of participants with change in nidus vascularity as assessed via MRI
Number of participants with changes in soft tissue and marrow edema as assessed via MRI | 12 months
  Number of participants with changes in soft tissue and marrow edema as assessed via MRI

CONTACTS AND LOCATIONS:
Overall Officials: Karun Sharma, MD, PhD, Principal Investigator — Children's National Research Institute
Locations (1):
- Children's National Hospital, Washington D.C., District of Columbia, United States

IPD SHARING:
Plan to Share IPD: No